CLINICAL TRIAL: NCT07117201
Title: Promoting Nutrition Security and Chronic Disease Management Through a Produce Prescription Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Ana Diallo, Assistant Professor, Virginia Commonwealth University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VCU HM20032577
Record Dates: First submitted 2025-06-30; First posted 2025-08-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Dietary Intervention; Produce Prescription; Chronic Disease Management; Social Needs Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Prescription Produce Program (PPP) (Active Comparator): The preliminary clinical effectiveness of the program on nutrition and food security status, diet quality as well as chronic disease management of individuals participating in the study
  Interventions: Behavioral: Prescription Produce Plan
- Standard Prescription Produce Program (PPP) + Cooking Classes (Experimental): The preliminary clinical effectiveness of the program on nutrition and food security status, diet quality as well as chronic disease management of individuals participating in the study AND cooking classes offered by Delicious Legacy.
  Interventions: Behavioral: Culturally Tailored Cooking Classes; Behavioral: Prescription Produce Plan

INTERVENTIONS:
Behavioral: Culturally Tailored Cooking Classes — Cooking skills session will be offered by the Delicious Legacy Program. The Delicious Legacy program is a culturally tailored, community-based nutrition and wellness intervention designed to promote health equity. Rooted in the intergenerational transmission of knowledge, the program emphasizes family socialization practices related to food, health beliefs, and caregiving. It integrates evidence-based nutritional education with ancestral foodways to address diet-related chronic illnesses while fostering cultural pride and resilience. Through interactive workshops, individuals engage in hands-on learning that reinforces traditional roles in food preparation and shared meals as sites of emotional support and identity formation.
  Arms: Standard Prescription Produce Program (PPP) + Cooking Classes
Behavioral: Prescription Produce Plan — The standard PPP includes three major parts. 1) Screening and personalized referrals/support for social needs including food, housing, health insurance and transportation by a community health worker. 2) Bi-weekly wellness visits with an MHWP team of interprofessional healthcare students, supervised by a clinical faculty, and guided by the participants' health and social needs and interests. They include education and SMART-EST goals around nutrition, physical activities, chronic disease management, care coordination, and/or recipes. 3) Delivery of a bag of fresh fruits and vegetables as well as heart healthy food items every two weeks over a period of 12 months. The produce bags will be made by the Underground Kitchen, a local non-profit organization creating curated bags of healthy food items and recipes to support the prevention and management of chronic diseases.

SUMMARY:
The goal of this study is to assess the feasibility to implement a prescription produce program (PPP) over 12-months within a community-based health and wellness program. The main questions it aims to answer are: a) does participation in the PPP improve participants' nutrition and food security status, health outcomes, diet quality and chronic disease management between baseline and 12 months after participating in the PPP? b) what is the cost-benefit analysis of the PPP implementation?

DETAILED DESCRIPTION:
Expanding the PPP over 12 months, incorporating additional healthy food items to increase variety, and including cooking skill sessions within the PPP will enhance participants' confidence in preventing and managing their chronic diseases. This initial assessment of the program will provide essential data for expansion and implementation. This PPP intervention will promote health equity by expanding the reach of our program and helping participants overcome SDOH, such as food insecurity, that prevent optimal diet quality and management of chronic diseases. Furthermore, continuous or more frequent monitoring of SDOH, provision of a variety of healthy food items, and lifestyle behavior change education should increase participant adherence to a more nutritious diet and medication management required for chronic disease management, and improve participants' chronic disease self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* a participant in the Mobile Health and Wellness Program;
* an English-speaking adult aged 18 or over
* diagnosed with hypertension, high cholesterol, diabetes type 2 or pre-diabetes, arthritis, obesity, CHF, and/or COPD
* taking medication for at least one of the eligible chronic conditions listed previously.

Exclusion Criteria:

* a prior diagnosis of dementia-related conditions: Alzheimer's disease, Lewy body, Parkinson's, or vascular dementia
* unwilling or unable to attend at least half of the 24 team visits during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in food security status at 12 months | From baseline to the end of intervention at 12 months
  The Hunger Vital Sign is a validated, two-question screening tool used to identify households at risk of food insecurity. It asks if within the past 12 months, the household has "worried whether our food would run out before we got money to buy more" or if "the food we bought just didn\'t last, and we didn\'t have money to get more". Answering that either statement is "often true" or "sometimes true" indicates a household is at risk.
Change in social needs | During active intervention from baseline to the end of study participation at 12 months
  The Social Needs Screening short survey will be used to measure social drivers of health, including housing, food insecurity, transportation, delayed care, and financial strain. Each domain is evaluated separately. A positive response is determined for each specific category (e.g., housing, food) rather than through a cumulative score.
Change from baseline in nutrition security status at 12 months | From baseline to the end of intervention at 12 months
  1-item Brief Nutrition Security Screener,
  Question: In the last 12 months, (I/we) worried that the food (I was/we were) able to eat would hurt (my/our) health and well-being.
  Response options:
  Always true Often true Sometimes true Never true Don't know / Refused Interpretation Responses of "Always true," "Often true," or "Sometimes true" typically indicate a level of nutrition insecurity.

SECONDARY OUTCOMES:
Change in hemoglobin A1c from baseline to 12 months | From baseline to end of study participation at 12 months
  Blood glucose level measured by hemoglobin A1c (HbA1c) levels using the DCA Vantage® Analyzer for individuals with diabetes and pre-diabetes
Change in diet quality from baseline to 12 months | From baseline to end of study participation at 12 months
  Dietary quality measured as the Healthy Eating Index using the DietID™, an assessment tool capturing dietary intake through an innovative Diet Quality Photo Navigation (DQPN®) software. Users are shown a series of food images representing different eating patterns and select the one that most closely resembles their own.The selected pattern is then evaluated using the HEI 2020 scoring system, a well-validated measure of how closely a diet aligns with the Dietary Guidelines for Americans. The HEI score (0-100) is converted into a simpler 1-10 scale, with 10 being the highest quality diet and 1 being the lowest.
Wellness goals set and completed during active study. | During active study engagement from baseline to end of study participation at 12 months
  Participants set a study-specific wellness goal related to lifestyle behaviors and chronic disease management at study baseline. Wellness goals are categorized by type of activity (e.g., physical activity, vegetable intake). During the MHWP team visits, participants will be supported to identify and design health and lifestyle behavior goals which will be SMART- EST (Specific, Measurable, Achievable, Relevant, Time-bound, Evidence-based, Strategic and Tailored). Participants provide progress updates and work towards optional action steps during visits through qualitative responses. Participants report if they achieved their wellness goal at study endpoint.
Change in global health from baseline to 12 months | From baseline to end of study participation at 12 months
  PROMIS Global Health includes global perceptions of general health that cut across physical and mental domains. The measure will assess the potential impact of the PPP on participants' overall health and chronic disease management. PROMIS Global Health scoring involves using the scores from specific health questions to calculate two summary scores: a Global Physical Health Score and a Global Mental Health Score. These scores are then standardized into "T-scores," where a score of 50 represents the average for the general population, with a standard deviation of 10
Change in food medication trade-offs from baseline to 12 months | From baseline to end of study participation at 12 months
  Food/medication trade-offs which will assess trade-offs between food and medications or diabetes supplies if they reported having a diagnosis of type 2 diabetes. We will use the following four Likert-scale questionnaire with response on 'often', 'sometimes', 'rarely' or 'never' to answer: "How often have you…:(1) put off buying food so that you would have money to buy medicines? (2) put off buying medicines so that you would have money to buy food? (3) put off buying diabetes supplies, like test strips or lancets, so that you would have money to buy food? (4) put off buying food so that you would have money to buy diabetes supplies, like test strips or lancets
Change in healthcare utilization | During active study participation from baseline to 12 months
  Self-reported healthcare utilization during team visits to include: last time seen at PCP, any hospitalizations or ER visits since last PPP visit or within the last month, # hospital and ER visits in last month, reasons for hospital and ER visits assessed during team visits. No standardized tool will be used.
Change in weight from baseline to 12 months | From baseline to end of study participation at 12 months
  Body weight measured using a calibrated digital scale
Change in adiposity from baseline to 12 months | From baseline to end of study participation at 12 months
  Adiposity which will be measured by waist circumference using the National Health and Nutrition Examination Survey protocol
Change in blood pressure from baseline to 12 months | From baseline to end of study participation at 12 months
  Blood pressure (SBP/DBP) measured by the Omron Hem 705 CP Auto Inflate BP Monitor
Change in medication adherence from baseline to 12 months | From baseline to end of study participation at 12 months
  Medication adherence will be measured using the Adherence to Refills and Medications Scale (ARMS) which assesses adherence with the filling or refilling of prescriptions, and adherence with taking medications. The Adherence to Refills and Medications Scale (ARMS) scoring involves summing the responses from its 12 items, each rated on a four-point scale (1 = none of the time, 4 = all of the time). Scores are then totaled to produce an overall score ranging from 12 to 48. A crucial part of the original scoring is a reverse coding of one item (usually item 12), meaning a higher score indicates poorer adherence, while a lower score indicates better adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Diallo, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Mobile Health and Wellness Program, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No